CLINICAL TRIAL: NCT02067806
Title: Observational Prospective Study on 2-chloroprocaine Hydrochloride 1% Safety in Intrathecal Anesthesia
Brief Title: Observational Study on 2-chloroprocaine Hydrochloride 1%
Acronym: PASS
Status: Completed | Type: Observational
Sponsor: Sintetica SA (Industry)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Other Study IDs: CHL1/01-2012/M
Record Dates: First submitted 2014-02-07; First posted 2014-02-20 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Neurological Complication, in Particular TNS or CES
Keywords: PASS; TNS; CES; CHLOROPROCAINE
MeSH Terms: conditions — Schmid-Fraccaro syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 2-chloroprocaine hydrochloride, 1% — Study included male and female adult patients undergoing spinal anesthesia with chloroprocaine, when the planned surgical procedure was not expected to exceeded 40 minutes.
  Other Names: Ampres 1%

SUMMARY:
The present study aims to evaluate the relationship between spinal block with 1% solution of 2-chloroprocaine hydrochloride and the onset of all possible neurological adverse events, with particular attention to Transient Neurological Symptoms (TNS) and Cauda Equina Syndrome (CES).

DETAILED DESCRIPTION:
Primary endpoint :Incidence of neurological complications (Transient and Permanent complications; e.g. transient neurological symptoms, arachnoiditis, cauda equina syndrome).Two follow-up questionnaires are foreseen, at 24 h and 7 days after time of spinal injection (Tsp), to gather all possible neurological complications, with particular attention to Transient Neurological Symptoms (TNS) and Cauda Equina Syndrome (CES).Patients scheduled for elective surgery will be informed about the aims, procedures and possible risks of the study and will be asked to sign the informed consent form for the inclusion in the trial, from day -14 to day of surgery (visit 1, Day 0).This observational study is planned to collect data on patients undergoing surgery under intrathecal anesthesia with chloroprocaine hydrochloride, primarily to assess the occurrence of all possible neurological adverse events (with particular attention to TNS and CES). The mandatory follow-ups of the study are at 24 h and 7 days (-1/+2) after anaesthesia. In case of signs of neurological complications, the patient has to undergo to a medical visit at the hospital by the relevant specialists (anaesthetist, surgeon, neurologist). In order to characterise the occurred adverse event, a complete analysis evaluation has to be conducted, as CT, MRI, Electromyography, etc. following the indication of the specialists. In case of persistent neuropathy the patient needs to be accurately followed according to the internal hospital procedure. In the meantime, a full screening of the patient's clinical history together with a detailed analysis of the relevant variables, potentially related to the adverse event, have to be carried out.

Therefore, the physician will take all appropriate measures to ensure the safety of the patients, notably he/she should follow up the outcome of any Adverse Events (clinical signs, laboratory values or other, etc.) until the return to normal or consolidation of the patient's condition. In case of any Serious Adverse Event, the patient has to be followed up until clinical recovery is complete and laboratory results have returned to normal, or until progression has been stabilized. The follow-up will continue after the patient has left the study.

ELIGIBILITY:
Inclusion Criteria:

* Male/female adult patients
* Ability to comprehend the full nature and purpose of the study
* Ability to co-operate with the Investigator and to comply with the requirements of the entire study
* Signed written informed consent of the patients prior to inclusion in the observational study. The signature has to be done before the elective surgery.
* Spinal anaesthesia in adults where the planned surgical procedure should not exceed 40 minutes.

Exclusion Criteria:

* Hypersensitivity to the active substance, medicinal products of the PABA (para-aminobenzoic acid) ester group, other ester-type local anaesthetics or to any of the excipients (Hydrochloric acid 1N for pH adjustment, Sodium chloride, Water for injection)
* General and specific contra-indications to spinal anaesthesia regardless of the local anaesthetic used, should be taken into account (e.g. decompensated cardiac insufficiency, hypovolemic shock….)
* Intravenous regional anaesthesia (the anesthetic agent is introduced into the limb and allowed to set in while tourniquets retain the agent within the desired area)
* Serious problems with cardiac conduction,
* Severe anaemia,
* It is also necessary to take into consideration general and specific contraindications for the technique of spinal anaesthesia = intrathecal anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery will be informed about the aims, procedures and possible risks of the study and will be asked to sign the informed consent form for the inclusion in the trial, from day -14 to day of surgery (visit 1, Day 0).
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2013-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Fanelli, MD, Principal Investigator — Azienda Ospedaliera di Parma Dipartimento di Anestesia, Rianimazione e Terapia Antalgica - Italy; Capdevila Xavier, MD, Principal Investigator — Head of the Department of Anesthesiology and Critical Care Medicine of Lapeyronie, France; Stefano Bonarelli, MD, Principal Investigator — Rizzoli Hospital, Bologna - Italy; John Van Delft, MD, Principal Investigator — Department of Anesthesiology and Critical Care Medicine, Belgium; Holger Sauer, MD, Principal Investigator — Klinik für Anästhesie, Intensivmedizin und Schmerztherapie; Martin Bauer, MD, Principal Investigator — Klinik für Anästhesiologie, Intensiv-, Palliativ- und Schmerzmedizin Berufsgenossenschaftliches; Laurent Delaunay, MD, Principal Investigator — Clinique générale d'Annency - La consultation d'Anesthésie
Locations (1):
- Department of Anesthesiology and Critical Care Medicine-Hospital AZ Sint Jozef, Malle, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Chloroprocaine 1%: Study included male and female adult patients undergoing spinal anesthesia with chloroprocaine, when the planned surgical procedure was not expected to exceeded 40 minutes.
Period: Overall Study
Arm/Group | Chloroprocaine 1%
Started | 394
Completed | 387
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- Chloroprocaine 1%: intrathecal anesthesia with 1% solution of 2-chloroprocaine hydrochloride in patients undergoing short surgical procedures (max. 40 minutes).
Arm/Group | Chloroprocaine 1%
Number analyzed (Participants) | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158
  Male | 235
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 388
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  Belgium | 200
  Germany | 139
  France | 54
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with neurological adverse events, with particular attention to Transient Neurological Symptoms (TNS) and Cauda Equina Syndrome(CES).
Time Frame: assessed at 24h and 7(-1/+2) days after surgery, total reported
Measure: Number; unit: participants
Arm/Group | Chloroprocaine 1%
Number analyzed (Participants) | 393
participants
  24 hours | 9
  7 days | 5

2. Primary Outcome: Number of Participants With Symptoms in Follow-Up Questionnaire at 24 Hours
Description: the follow-up questionnaires are foreseen, at 24 h after time of spinal injection (Tsp), to gather all possible neurological adverse events. About 24 h after surgery (indicated as Tsp),Investigator or a deputy will question patients about neurological symptoms and pain not associated to the operation area on the basis of the follow-up questionnaires and giving a score between 0 to 10 to the pain intensity. All other adverse events will also be assessed.
Time Frame: 24 hours
Measure: Number; unit: number of patients
Arm/Group | Chloroprocaine 1%
Number analyzed (Participants) | 393
number of patients
  fatigue | 4
  nausea/vomiting | 3
  dizziness | 1
  urin/defec problems | 1

3. Primary Outcome: Number of Participants With Symptoms in Follow-Up Questionnaire at 7 Days
Description: the follow-up questionnaires are foreseen, at 7 days after time of spinal injection (Tsp), to gather all possible neurological adverse events. About 7 days after surgery (indicated as Tsp),Investigator or a deputy will question patients about neurological symptoms and pain not associated to the operation area on the basis of the follow-up questionnaires and giving a score between 0 to 10 to the pain intensity. All other adverse events will also be assessed.
Time Frame: 7 days
Measure: Number; unit: number of patients
Arm/Group | Chloroprocaine 1%
Number analyzed (Participants) | 393
number of patients
  fatigue | 3
  nausea/vomiting | 1
  dizziness | 1
  urin/defec problems | 2

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Chloroprocaine 1%
All-Cause Mortality (participants affected / at risk) | 0/393
Serious Adverse Events (participants affected / at risk) | 0/393
Other Adverse Events (participants affected / at risk) | 37/393
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroprocaine 1% (N=393)
bradycardia (Cardiac disorders) | 4 (4)
vomiting (Gastrointestinal disorders) | 2 (2)
drug effect incomplete (General disorders) | 4 (4)
drug ineffective (General disorders) | 1 (1)
injection site pain (General disorders) | 1 (1)
anesthetic complication (Injury, poisoning and procedural complications) | 3 (3)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 6 (6)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
burning sensation (Nervous system disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2)
hypotonia (Nervous system disorders) | 2 (2)
paresthesia (Nervous system disorders) | 4 (4)
hyprventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypotension (Vascular disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No